CLINICAL TRIAL: NCT00935597
Title: A Phase I Trial of Host Dendritic Cell Infusion After Allogeneic Stem Cell Transplant for Prevention or for Treatment of Relapsed Disease in Patients With Advanced Hematologic Malignancies
Brief Title: Host Dendritic Cells in Allograft Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Keren Osman, MD, Principal Investigator, Mount Sinai School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-0906
Record Dates: First submitted 2009-07-07; First posted 2009-07-09 (Estimated); Last update posted 2010-10-29 (Estimated); Status verified 2010-10

CONDITIONS: Relapsed Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma; Chronic Lymphocytic Lymphoma
Keywords: Relapsed Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma; Chronic Lymphocytic Lymphoma; Relapsed Non-Hodgkin's lymphoma (excluding follicular lymphoma and marginal zone lymphoma)
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Lymphoma, B-Cell, Marginal Zone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Patients with Minimal Residual Disease or Minimal Volume Relapse post allogeneic stem cell transplant will receive MSSM/BIIR HDC Vax-001 (Host Dendritic Cells) by infusion
  Interventions: Biological: MSSM/BIIR HDC Vax-001 (Host Dendritic Cells)
- Group 2 (Experimental): Patients with greater than Minimal Residual Disease or Minimal Volume Relapse post allogeneic stem cell transplant will receive MSSM/BIIR HDC Vax-001 (Host Dendritic Cells) by infusion in conjunction with donor lymphocyte infusion (DLI)
  Interventions: Biological: MSSM/BIIR HDC Vax-001 (Host Dendritic Cells)

INTERVENTIONS:
Biological: MSSM/BIIR HDC Vax-001 (Host Dendritic Cells) — Patients who have minimal residual disease or minimal volume relapse, and are at least four weeks post immunosuppression following allogeneic stem cell transplantation will receive a series of four HDC infusions (100,000 HDC/kg per infusion, one every four weeks(group 1). Those patients who have greater than minimal residual disease will receive HDC infusions, one every four weeks in conjunction with donor lymphocyte infusion (DLI) (group 2).

SUMMARY:
The purpose of this study is to assess preliminary efficacy and to determine the safety and feasibility of ex vivo generated dendritic cell (HDC) infusion with and without donor lymphocyte infusion (DLI) after allogeneic stem cell transplant (SCT). We also wish to establish the feasibility of apheresis shipment as well as vaccine shipment and stability in the population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70
* Ability to sign informed consent
* ECOG performance status ≤3
* Life expectancy > 6 months
* Adequate cardiac function: MUGA or Echocardiogram demonstrating >50% Ejection Fraction
* Adequate pulmonary function with DLCO > 50%
* Adequate hepatic function

  * Bilirubin ≤ 1.5mg/dl
  * Alkaline phosphatase ≤5 times the upper limit of normal
  * Aspartate aminotransferase (AST) or serum glutamic-oxaloacetic transferase (SGOT) ≤ 3 times the upper limit of normal
  * Alanine aminotransferase (ALT) or serum glutamic pyruvic transaminase (SGPT) ≤ 3 times the upper limit of normal
* Adequate renal function Estimated creatinine clearance > 40ml/min
* Diagnosis of one of the following

  * Non-Hodgkin's lymphoma excluding Follicular lymphoma and Marginal Zone Lymphoma
  * Hodgkin's lymphoma
  * Multiple myeloma
  * Chronic lymphocytic leukemia
* Eligible for allogeneic stem cell transplant with identified HLA-identical sibling (6/6 HLA match) or volunteer unrelated donor (8/8 allele HLA-matched (A, B, Cw, DRB1)
* Women of childbearing potential must have a negative serum pregnancy test prior to enrollment
* Women of childbearing potential must use effective means of birth control throughout the study.
* Men should not father a child while enrolled in the study. Effective means of birth control include condom, vasectomy or abstinence.

Exclusion Criteria:

* Malignancies other than melanoma within five years of study entry, except carcinoma in-situ of the cervix or basal/squamous cell skin cancers
* Concurrent illnesses that would preclude survival > 6 months other than the disease under study
* Pregnancy or nursing
* HIV infection
* Treatment with prior donor lymphocyte infusion
* Prior allogeneic stem cell transplant
* History of autoimmune diseases including systemic lupus erythematosus, rheumatoid arthritis and thyroiditis
* Active infections including fungal infections and viral hepatitis
* GVHD greater than grade I GVHD of the skin

Patient Exclusion Criteria for Part B (post Stem Cell Transplant)

* Malignancies other than melanoma within five years of study entry, except carcinoma in-situ of the cervix or basal/squamous cell skin cancers
* Concurrent illnesses that would preclude survival > 6 months other than the disease under study.
* Pregnancy or nursing
* HIV infection
* Treatment with prior donor lymphocyte infusion
* Prior allogeneic stem cell transplant
* More than 4 prior relapses
* History of autoimmune diseases including systemic lupus erythematosus, rheumatoid arthritis and thyroiditis
* Active infections including fungal infections and viral hepatitis
* GVHD greater than grade I GVHD of the skin
* No cytotoxics will be given within 4 weeks of administration of the investigational cell therapy
* Patients cannot receive any investigational agents within 30 days prior to administration of the investigational cell therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
The incidence of severe graft versus host disease (GVHD) grade C or D as defined by IBMTR grading. | 2 weeks following each HDC infusion and 4, 6 and 8 weeks after the last HDC infusion

SECONDARY OUTCOMES:
The incidence of grade A and B acute GVHD, limited chronic GVHD, infusion reactions, graft loss and donor chimerism | 2 weeks following each HDC infusion and 4, 6 and 8 weeks after the last HDC infusion

CONTACTS AND LOCATIONS:
Overall Officials: Keren Osman, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States